CLINICAL TRIAL: NCT03831282
Title: Feasibility and Performance Evaluation of INVSENSOR00024
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHOC0004
Record Dates: First submitted 2019-02-04; First posted 2019-02-05 (Actual); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Evaluation of SpO2 Performance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- RD SET Neo SpO2 (Experimental): All subjects enrolled in the study will receive the investigational sensor (RD SET Neo SpO2) for evaluation of SpO2.
  Interventions: Device: RD SET Neo SpO2

INTERVENTIONS:
Device: RD SET Neo SpO2 — All subjects are enrolled in the experimental group and receive the RD SET Neo SpO2 sensor.

SUMMARY:
This is a prospective, non-randomized, single arm study design to evaluate SpO2 performance of the INVSENSOR00024 sensors in the neonatal population in a clinical environment using convenience sampling.

ELIGIBILITY:
Inclusion Criteria:

* Less than or equal to 1 month (28 days) of age
* Weight ≤ 5 kg at the time of consent or last recorded weight prior to consent.
* Subjects admitted with standard of care (SOC) arterial blood sampling line already in place

Exclusion Criteria:

* Subjects with both significant abnormal aortic arch and radial line in place
* Subjects with suspected or diagnosed critical congenital heart disease (CCHD)
* Subjects with underdeveloped skin
* Subjects with abnormalities at the planned application sites that would interfere with system measurements
* Subjects with known allergic reactions to foam/rubber products and adhesive tape
* Deformities of limbs, absence of feet, severe edema, and other at the discretion of the Principal Investigator

Max Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RD SET Neo SpO2
Started | 12
Completed | 11
Not Completed | 1
Not completed — Could not place sensor | 1

BASELINE CHARACTERISTICS:
Arm/Group | RD SET Neo SpO2
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Oxygen Saturation (SpO2) Measurement by RMS Calculation
Description: Accuracy will be determined by comparing the noninvasive blood oxygen saturation measurement of the pulse oximeter to that obtained from a blood sample and calculating the root mean square (RMS) error value. In order to obtain the RMS value, the blood oxygen saturation measurement form a laboratory pulse Co-Oximeter is subtracted from the pulse oximeter oxygen saturation measurement for each sample, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the RMS Error value.
Time Frame: up to 12 hours
Population: Subject 5:Removed per ISO standard for SpO2 equal to 100. Subject 12: No data collected
Measure: Number; unit: percent of oxygen saturated hemoglobin
Arm/Group | RD SET Neo SpO2
Number analyzed (Participants) | 10
percent of oxygen saturated hemoglobin | 3.5

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | RD SET Neo SpO2
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT03831282/Prot_SAP_000.pdf